CLINICAL TRIAL: NCT06814925
Title: Italian Prospective Observational Cohort Study of Patients With Lymphoma
Brief Title: Italian Study of Patients With Lymphoma
Acronym: LYMPH-OS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: LYMPH-OS
Record Dates: First submitted 2024-12-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma
Keywords: questionnaire
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
It is an observational, non-interventional, prospective, monocentric study, whose objective is to enroll 1500 patients with lymphoma in 5 years within the Institute of Hematology "Seragnoli".

DETAILED DESCRIPTION:
The study is aimed at enriching the data on the prognostic role of genetic and epidemiological factors associated with clinical and epidemiological data of patients; to identify factors that influence the evolution of the disease, such as lifestyle and occupational factors, as well as the type of treatment; to document the impact of the disease on quality of life and to provide a platform for future research projects.

Study-specific questionnaires will be administered to patients, both at baseline and during follow-up, which methodologically represent a useful tool in order to achieve these objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at enrollment
* Diagnosis of lymphoma within 3 months of enrollment
* Patients may have been treated, as long as the initial diagnosis of lymphoma is within 3 months of enrollment
* Signing of the informed consent form

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1500 patients with lymphoma (about 500 cases of DLBCL, 360 of FL, 260 of CLL/SLL, 110 of MZL, 60 of PTCL e MCL, 40 of LPL/WM, 30 of MF and BL, and 15 of HCL e ALL)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 5 years
  From the date of diagnosis to the date of death

SECONDARY OUTCOMES:
Event Free Survival (EFS) | through study completion, an average of 5 years
  Time elapsed from the date of diagnosis to the date of the first event that occurred (disease progression, relapse or new treatment for lymphoma, or death)
Lymphoma Specific Survival (LSS) | through study completion, an average of 5 years
  Time elapsed from the date of diagnosis to the date of death from lymphoma (disease progression, relapse or new treatment for lymphoma, or death)
Progression-Free Survival (PFS) | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
net survival | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
response rate | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Duration of response | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Time to next anti-lymphoma treatment (TTNLT) | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Duration of survival after progression | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Frequency of lymphoma transformation | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Frequency of secondary cancers | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
Frequency of other chronic diseases | through study completion, an average of 5 years
  To enrich data on the prognostic role of associated genetic and epidemiological factors with clinical and epidemiological data from patients and to identify factors affecting disease progression, such as lifestyle and occupational factors, as well as the type of treatment
questionnarire of Quality of Life FACT-LYM (Functional Assessment of Cancer Therapy-Lymphoma): score 0 to 4 | through study completion, an average of 5 years
  questionnarire of Quality of Life FACT-LYM (Functional Assessment of Cancer Therapy-Lymphoma): score 0 to 4.questions regarding physical well-being, social/familial well-being, emotional well-being, functional well-being, additional questions specific to lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No